CLINICAL TRIAL: NCT02114333
Title: A Comparison of the Immunogenicity and Descriptive Safety of a Live Attenuated Herpes Zoster Vaccine and the Glaxo Smith Kline (GSK) Herpes Zoster Recombinant HZ/su Candidate Vaccine in 50-59 Year Old and 70-85 Year Old Vaccine Recipients
Brief Title: Comparison of a Live Herpes Zoster Vaccine and a Recombinant Vaccine in 50-59 and 70-85 Year Olds
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 13-3192
Record Dates: First submitted 2014-04-11; First posted 2014-04-15 (Estimated); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Shingles; Herpes Zoster
Keywords: Shingles vaccine; Immune response; Zoster vaccine
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Vaccines, Synthetic; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

ARMS (4):
- A - Live zoster vaccine (Active Comparator): No previous zoster vaccine; stratified between age groups 50-59 and 70-85
  First dose live vaccine, Zostavax (0.65ml, subcutaneous)
  Second dose placebo, normal saline (0.65ml. subcutaneous)
  Interventions: Biological: Zostavax; Biological: Placebo
- B - recombinant zoster vaccine (Active Comparator): No previous zoster vaccine; stratified between age groups 50-59 and 70-85
  First dose recombinant vaccine, HZ/su (0.5ml, intramuscular)
  Second dose recombinant vaccine, HZ/su (0.5ml, intramuscular)
  Interventions: Biological: HZ/su vaccine
- C - Live zoster vaccine (Active Comparator): One previous dose of zoster vaccine at least 5 years previously, age 70-85
  First dose live vaccine, Zostavax (0.65ml, subcutaneous)
  Second dose placebo, normal saline (0.65ml. subcutaneous)
  Interventions: Biological: Zostavax; Biological: Placebo
- D - recombinant zoster vaccine (Active Comparator): One previous dose of zoster vaccine at least 5 years previously, age 70-85
  First dose recombinant vaccine, HZ/su (0.5ml, intramuscular)
  Second dose recombinant vaccine, HZ/su (0.5ml, intramuscular)
  Interventions: Biological: HZ/su vaccine

INTERVENTIONS:
Biological: Zostavax — 0.65ml, subcutaneous
  Arms: A - Live zoster vaccine; C - Live zoster vaccine
Biological: HZ/su vaccine — 0.5ml, intramuscular
  Other Names: Recombinant vaccine
  Arms: B - recombinant zoster vaccine; D - recombinant zoster vaccine
Biological: Placebo — 0.65ml, subcutaneous
  Other Names: normal saline
  Arms: A - Live zoster vaccine; C - Live zoster vaccine

SUMMARY:
This study will compare the two vaccines that have been developed to prevent and/or lessen the effects of shingles. One vaccine is live (Zostavax, licensed by FDA) and the other, herpes zoster subunit (HZ/su), contains a piece of the shingles virus (not live) and an ingredient that may enhance the body's immune response to the vaccine, and is currently investigational. The vaccines are being compared to assess their ability to stimulated protection against shingles. The study will provide an opportunity to determine the safety profile of each vaccine in a single trial. The study will also look at the effect of age on the immune response to the two vaccines and on the persistence of these responses.

DETAILED DESCRIPTION:
160 people from the Denver area will participate. Duration is up to 5 years with 10-12 visits in that period. Subjects are randomized into one of 4 arms to receive either Zostavax or HZ/su. In this single blind study all subjects receive 2 injections: one at the first visit (Day 0) and the second at Day 60. HZ/su subjects will receive vaccine at both visits; Zostavax subjects will receive vaccine at the first visit and a placebo at the Day 60 visit. Blood is collected from all subjects at most visits. Some subjects spit into a tube for saliva collection. A urine sample is collected prior to vaccination if subject is a woman of childbearing potential. Subjects are asked to complete a diary to record any reactions in the 30 days after each injection. The Day 90 visit is the last one until the annual visits for blood draws begin at Day 365. Some subjects are also seen at Year 2 and Year 4; all subjects are seen at Year 5 for blood draw.

ELIGIBILITY:
Inclusion Criteria:

* History of varicella or residence int he US for 30 years
* For Arms C and D - prior live zoster vaccine at least 5 years previously
* For Arms A and B - Age 50-59 or 70-85
* For Arms C and D - Age 70-85
* For women of childbearing potential, a negative pregnancy test and agreement to use adequate contraception from 30 days before until 3 months after the last dose of any study vaccine

Exclusion Criteria:

* History of herpes zoster
* For Arms A and B - prior live zoster vaccine
* Immune compromising illness or therapies or chronic illness
* Allergy to previous herpes zoster vaccine
* Other investigational drugs or vaccines within the past 6 months before the study and until last visit
* Blood products for 3 months prior to or planned during the study
* Concomitant non-topical antiviral therapy within 3 days prior to and 7 days after vaccination.
* Vaccines within 2 weeks (inactive vaccine) or 4 weeks (live vaccine) prior to the study until 30 days after any dose of either vaccine.
* Pregnancy or breast-feeding
* Current drug addiction or alcoholism.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2020-05 (Actual)

PRIMARY OUTCOMES:
Changes in Interferon gamma/ Interleukin 2 (IFNg/IL2) dual color fluorospot number | Measured up to Day 730

SECONDARY OUTCOMES:
Changes in glycoprotein-based enzyme-linked immunosorbent assay (gpELISA) | Measured up to Day 730

OTHER OUTCOMES:
Evaluation of Unsolicited adverse events | Within 30 days of each vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Myron J Levin, M.D., Principal Investigator — University of Colorado School of Medicine
Locations (1):
- Pediatric Infectious Diseases and Clinical Trials, Universtiy of Colorado School of Medicine, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Johnson MJ, Liu C, Ghosh D, Lang N, Levin MJ, Weinberg A. Cell-Mediated Immune Responses After Administration of the Live or the Recombinant Zoster Vaccine: 5-Year Persistence. J Infect Dis. 2022 Apr 19;225(8):1477-1481. doi: 10.1093/infdis/jiab580. PMID 34850039
- [Derived] Weinberg A, Kroehl ME, Johnson MJ, Hammes A, Reinhold D, Lang N, Levin MJ. Comparative Immune Responses to Licensed Herpes Zoster Vaccines. J Infect Dis. 2018 Sep 22;218(suppl_2):S81-S87. doi: 10.1093/infdis/jiy383. PMID 30247596